CLINICAL TRIAL: NCT03752125
Title: A Randomized, Cross-Over Clinical Trial to Evaluate the Acute Effects of Mixed Flavonoid and Caffeine Ingestion on Energy Expenditure and Fat Oxidation in Healthy Adult Women
Brief Title: Influence of Flavonoids and Caffeine Supplementation on Resting Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 18-0257
Record Dates: First submitted 2018-05-03; First posted 2018-11-23 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Diet Modification
Keywords: energy expenditure; caffeine; flavonoids; fat metabolism
MeSH Terms: interventions — Flavonoids; Caffeine

STUDY DESIGN:
Intervention Model Description: Randomized, crossover
Who Masked: Participant, Investigator
Masking Description: Flavonoid and placebo capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flavonoid, caffeine (Experimental): Flavonoid, caffeine capsules
  Interventions: Dietary Supplement: Flavonoid, caffeine
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Flavonoid, caffeine — 2 flavonoid/caffeine capsules before breakfast, 2 capsules before lunch
  Arms: Flavonoid, caffeine
Dietary Supplement: Placebo — 2 placebo capsules before breakfast, 2 capsules before lunch
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effect of ingesting caffeine and mixed flavonoids (4 capsules, split between breakfast and lunch) on energy expenditure and fat oxidation in a metabolic chamber with 20 women (non-obese, healthy, ages 20-47 years, pre-menopausal). We hypothesize that based on the existing literature, ingestion of a double dose of the caffeine-mixed flavonoid supplement compared to placebo will increase fat oxidation and increase 24 h energy expenditure by about 75 kilocalories.

DETAILED DESCRIPTION:
This study will utilize a randomized, double-blind, cross-over design, comparing acute ingestion of the mixed flavonoid supplement (MF) compared to placebo control (PC) in healthy, non-obese, pre-menopausal women. The study will consist of two 24-hour study periods spent in the recently renovated indirect room calorimeter (i.e., metabolic chamber) at the University of North Carolina Chapel Hill Nutrition Research Institute (UNC NRI). The 24-hour study periods in the metabolic chamber will be 4 weeks apart. Primary outcome measures will be 24-hour energy expenditure (EE), resting metabolic rate (RMR), sleeping metabolic rate (SMR), substrate utilization from the respiratory quotient (RQ), and physical activity energy expenditure (AEE).

Following recruitment and eligibility assessment, study participants will be randomly assigned to complete either the mixed flavonoid (MF) or the placebo control (PC) study day. After a 4-week washout, study participants will cross over and complete the alternative treatment. A method of randomly permuted blocks will be generated using web-based randomization software (www.randomization.com) resulting in 10 study participants receiving MF during the first week, and 10 study participants receiving the PC during the first week. Study participants will consume 2 MF or PC capsules 30 min before breakfast, and 2 MF or PC capsules 30 min before lunch. During both study days, study participants will be fed in energy balance (i.e., energy intake will be matched to energy expenditure).

2. Experimental Study Participants: Using data generated previously in the UNC NRI metabolic chamber, a sample size calculation with 80% power revealed that 15-20 study participants would be needed to detect a 50 kcal difference in 24-h EE. To account for attrition, 25 study participants will be recruited via mass advertisement throughout the local area. Pre-menopausal women will be chosen because this is a target population of the sponsor.

3. Pre-Study Baseline Testing Eligibility will be determined in the outpatient clinical suite at the UNC NRI. Body composition (fat mass and fat free mass (FFM)) will be determined via dual energy x-ray absorptiometry (DXA) (GE Lunar iDXA; Milwaukee, WI). Body mass index (BMI, kg/m2) will be calculated for measured height and weight. Resting metabolic rate (RMR) will be estimated using a FFM-based equation [418 + (20.3 FFM)] (J Appl Physiol 1993;75:2514-2520). This estimated RMR will be used to calculate total dietary energy intake while in the metabolic chamber: RMR x physical activity level (PAL) of 1.3, and then adjusted using measured data (details provided below). A small blood sample will be obtained at this time and T3, T4, and TSH levels assessed through the clinical lab at the Lab Corp (Burlington, NC). A urine pregnancy test will be performed.

4. Indirect calorimetry: The metabolic chamber at the Nutrition Research Institute in Kannapolis, NC is an open-circuit, whole room indirect calorimeter. The CO2 and O2 analysers are differential, with full scale readings set for 0%-1%. O2 consumption, CO2 production, EE and RQ are recorded each minute. EE is calculated using an abbreviated Weir's formula (VO2 X 3.941) + (VCO2 X 1.106), where VO2 is the volume of oxygen consumed in L/minute and VCO2 is the volume of carbon dioxide released in L/minute. RQ is calculated as VCO2/VO2. Area under the curve (AUC) will be calculated using RQ data for the four hours following breakfast, lunch and dinner as well as sleeping hours between midnight and 6:00 am. Spontaneous physical activity will be measured each minute using a total room sensor. To calculate resting metabolic rate (RMR), EE will be plotted against the activity motion sensor output (each averaged over 30 minutes), and the y-intercept of the linear regression taken as EE in the inactive state. RMR will be multiplied by 1440 minutes to extrapolate to 24 hours. Twenty-four hour sleeping metabolic rate (SMR) will be determined as the lowest mean EE (kJ/minute) measured over 3 consecutive hours between midnight and 6:30 am and multiplied by 1440 minutes. Diet induced thermogenesis (DIT) will be calculated by subtraction of SMR from RMR. Activity induced EE (AEE) will be calculated as the difference between 24 hour EE and RMR.

5. Metabolic chamber study day protocol. Subjects will arrive at the Nutrition Research Institute Building (500 Laureate Way) at 7:00 am. A urine pregnancy test will be performed. At 7:30 am, study participants will report to the metabolic chamber following an overnight fast (no food or beverages containing calories, alcohol, or caffeine from 11 pm). Study participants will be instructed on expectations of their stay and weighed in scrubs without shoes. At 8:00 am study participants will be sealed in the chamber. Except for a 2-minute interval each hour during which study participants will be requested to stand and stretch, study participants will remain seated or reclined, but awake throughout the day. Study participants will be asked to perform necessary daily activities during these 2-minute intervals. Breakfast (9:00 am), lunch (1:30 pm), and dinner (7:00 pm), will be served through an air-lock passage. Meals will be completed within 30 minutes of serving. Two MF capsules or placebo will be consumed 30 min before breakfast, and then again 30 minutes before lunch. At 10:30 pm, study participants will be asked to lie down for sleep. Study participants will be awakened at 6:30 am and allowed to move about the chamber to gather their belongings. At 7:15 am study participants will exit the chamber and be weighed.

6. Design of Metabolic Diets: Eucaloric diets will be designed to provide approximately 35% fat, 49% carbohydrates and 16% protein, reflecting current recommendations for this population group. Menus will be designed using a nutrient calculation and food management software, and consist of bagel, peanut butter, apple juice, whole-wheat bread, turkey, cheese, mayonnaise, buttery spread (10% kcal as fat), potato chips, lasagna, carrots, broccoli, rolls, and muffin. No beverages or foods containing caffeine will be served. The same foods will be served at both chamber visits. A baseline menu for each subject will be prepared based on calculated RMR X 1.3, reflecting the sedentary nature of the study day. To ensure energy balance conditions, the baseline menu of the first visit will be modified according to measured EE data at 3 hours (includes breakfast) and 7 hours (includes breakfast and lunch). Subsequent meals will be adjusted accordingly with 100 kcal peach muffins containing the same proportion of fat, carbohydrate and protein as the meals. Study participants will be fed an identical amount of the same meal at their second visit.

7. Statistical Analysis: Data will be analyzed using SAS (Cary, NC). To guard against any carryover effect from visit 1 to visit 2, a repeated measures regression with an unstructured correlation matrix within subject will be run with treatment (MF and PC) and visit (1 and 2) in the model along with an interaction term. If the interaction term is non-significant, then it will be removed and the model re-run. Two energy expenditure curves, one for the MF day, and one for the PC day, will be generated for each subject with the x axis representing time (min), and the y axis representing energy expenditure (kcal). The area under the energy expenditure curve for defined blocks of time will be calculated by using the trapezoid rule in the EXPAND procedure in SAS (SAS Institute, Inc., Cary, NC). A paired t-test on the log-transformed area will be performed to compare the energy expenditure of each period in the MF day with the corresponding period in the PC day. The Shapiro-Wilk test in the UNIVARIATE procedure in SAS will be used for normality check. The Benjamini-Hochberg method for false discovery rate correction in the MULTTEST procedure in SAS will be used for multiple testing corrections.

SUPPLEMENT:

The mixed flavonoid supplement and placebo capsules will look identical and be supplied by Reoxcyn Discoveries Group LLC (Salt Lake City, UT). Active ingredients in the flavonoid capsules include vitamin C, wild bilberry fruit extract, green tea leaf extract, quercetin, caffeine, and omega 3 fatty acids (see Appendix B). Capsule fill ingredients include Nu-Flow 70R (from powdered rice hulls), tapioca from cassava root, natural bamboo silica, and marshmallow root. Placebo capsules will contain only the fill ingredients (without the active ingredients). Two MF and PC capsules will be consumed 30 minutes before breakfast, and then again before lunch. The MF capsules will provide 658 mg flavonoids and 214 mg caffeine.

ELIGIBILITY:
Inclusion Criteria:

* Women, ages 20 to 47 years
* Body mass index (BMI) between 18.5 and 33 kg/m2 (normal weight, overweight, mild obesity)
* Weight during the past 6 months has been somewhat stable (+/- 12 lbs)
* Low-to-moderate caffeine intake, defined as consuming on average: less than 3 servings per day of coffee (each about 8 fl. oz.) and/or energy drinks with caffeine; less than 3 soft drinks with caffeine and tea per day
* Premenopausal (self-report)
* Willingness to maintain habitual diet and physical activity patterns, and not lose weight throughout the study period
* Understands and agrees to all study procedures and signs the form providing informed consent to participate in the study
* Willingness to report and maintain normal schedule of hormonal therapy including oral contraceptive pills, hormonal IUD, Nuva Ring, or DepoProvera injections.
* Normal thyroid function as determined from a blood sample collected during pre-study baseline testing.
* Not pregnant as determined by a urine pregnancy test during pre-study baseline testing and prior to the second chamber session, and not planning to become pregnant during the study.
* Willingness to avoid vigorous exercise the day before each metabolic chamber session (e.g., intense running, cycling, swimming for 30 minutes and longer).

Exclusion Criteria:

* Taking medications for or suffering from a medical condition that may impact results related to metabolism (e.g. thyroid disorders, diabetes, mental disorders such as anxiety or depression, heart disease, arthritis, cancer).
* Heavy exerciser (defined as more than 300 minutes per week of moderate to vigorous exercise within the last two weeks)
* Thyroid hormone levels outside of the normal laboratory reference range
* Pregnant or lactating, or planning to become pregnant during the study
* Recent use of antibiotics (within last two weeks)
* History of smoking during the six months prior to study
* Recent signs or symptoms of infection, including cold or flu-like symptoms (within last 2 weeks)
* Conditions or diseases the investigator believes would interfere with ability to provide consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk. These include the disease list above and other health problems that would make it difficult to comply with two 24-hour periods of confinement in the metabolic chamber such as panic disorder, cardiac arrhythmias, musculoskeletal disorders such as low back pain and osteoarthritis, and gastrointestinal disorders including reactions to supplements with caffeine and vitamin C, and food allergies.
* Inability or unwillingness to consume the foods that will be included in the provided meals when staying in the chamber
* History of drug or alcohol abuse (>5 standard drinks per day)
* Taking herbal supplements or medications that may influence metabolism within 14 days prior to the study, including supplements containing bitter orange, guarana, fucoxanthin, and green coffee bean, and medications such as Meridia, Xenical, LipoRidAM, Advantra-Z, NuPhedrine, and Slim-10.
* Current consumption (or unwilling to stop intake 2 weeks prior) of flavonoid supplements, or a heavy consumer of green tea (>3 cups per day)
* Near-daily use of tablets containing caffeine (e.g., NoDoz) (or unwillingness to stop 2 weeks prior to the study).
* High intake of caffeine from coffee, tea, energy drinks with caffeine, and soft drinks containing caffeine (or unwillingness to reduce intake for 2 weeks prior to the study and during the 4-week study).
* Prone to panic attacks when confined in a small room, especially when consuming caffeine.

Ages: 20 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 25 (Actual)
Dates: Start 2018-04-22 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
24-hour energy expenditure (kilocalories/minute) from continuous respiratory exchange measurements (oxygen consumption, carbon dioxide production) in a metabolic chamber | 24 hours
  Energy expenditure (kilocalories) over 24 h in metabolic chamber with oxygen consumption and carbon dioxide production analyzers whereby energy expenditure is calculated from respiratory exchange data (oxygen consumption, carbon dioxide production) using standard equations

SECONDARY OUTCOMES:
24-hour fat oxidation (fat grams oxidized per minute) from continuous respiratory exchange measurements (oxygen consumption, carbon dioxide production) in a metabolic chamber | 24 hours
  Fat oxidation (fat grams) over 24 h in metabolic chamber with oxygen consumption and carboh dioxide production analyzers whereby fat oxidation (grams/minute) is calculated from respiratory exchange data (oxygen consumption, carbon dioxide production) using standard equations

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State Univ
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No